CLINICAL TRIAL: NCT01814722
Title: Quality of Life of HIV-infected Patients Switched to Raltegravir Versus Other Antiretroviral Regimens
Brief Title: Quality of Life of HIV-infected Participants Switched to Raltegravir Versus Other Antiretroviral Regimens (MK-0518-266)
Status: Terminated | Type: Observational
Why Stopped: The trial was terminated early due to slow recruitment.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0518-266
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV Infections; Anti-HIV Agents; Anti-Retroviral Agents; Nucleoside Reverse Transcriptase Inhibitors; Non-nucleoside Reverse Transcriptase Inhibitor; Protease inhibitors
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Raltegravir + 2 NRTIs: Raltegravir is an integrase inhibitor. Two Nucleoside Reverse Transcriptase Inhibitor (NRTIs)
- NNRTI + 2 NRTIs: Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI) could include: delavirdine, efavirenz, etravirine, rilpivirine, nevirapine; and two NRTIs.
- PI + 2 NRTIs: Protease inhibitors (PI) could include: nelfinavir, lopinavir, saquinavir, tipranavir, atazanavir and darunavir; and two NRTIs.

SUMMARY:
This is a multi-center, longitudinal observational study of adult human immunodeficiency virus (HIV) participants at academic and community-based practices in the United States who are switching from first-line to second-line therapy. The study's primary hypothesis is that HIV participants switching to raltegravir-based regimens will have better Medical Outcomes Study-HIV (MOS-HIV) Health Survey scores than participants switched to non-nucleoside reverse transcriptase inhibitor (NNRTI)-based or protease inhibitor (PI)-based regimens.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV
* Switching antiretroviral regimen(s) for the first time at the start of the study

Exclusion Criteria:

* Currently pregnant
* Presence of active tuberculosis, Hepatitis B, and/or Hepatitis C and receiving treatment for the condition(s) during the study period
* Presence of active pneumonia or other signs of opportunistic infections at the start of the study
* Currently participating in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients at academic and community-based practices in the United States
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-11-09 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0518-266&kw=0518-266&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with human immunodeficiency virus (HIV) who were switching from first-line antiretroviral regimens to a second-line regimen were recruited at 48 academic and community-based practices in the U.S.A.
Groups:
- Raltegravir + 2 NRTIs: Participants were treated with raltegravir (an integrase inhibitor), and two nucleoside reverse transcriptase inhibitors (NRTIs)
- NNRTI + 2 NRTIs: Participants were treated with two NRTIs and a non-nucleoside reverse transcriptase inhibitor (NNRTI).
- PI + 2 NRTIs: Participants were treated with two NRTIs and a protease inhibitor (PI).
Period: Overall Study
Arm/Group | Raltegravir + 2 NRTIs | NNRTI + 2 NRTIs | PI + 2 NRTIs
Started | 36 | 21 | 6
Completed | 36 | 21 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Gender and Age data for one participant from the Raltegravir, and two participants from the NNRTI groups were missing, resulting in a n = 60.
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir + 2 NRTIs | NNRTI + 2 NRTIs | PI + 2 NRTIs | Total
Number analyzed (Participants) | 35 | 19 | 6 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.7 (8.9) | 45.2 (13.8) | 48.8 (4.1) | 46.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 2 | 0 | 16
  Male | 21 | 17 | 6 | 44

OUTCOME MEASURES:

1. Primary Outcome: Medical Outcomes Study-HIV (MOS-HIV) Health Survey Scores
Description: The MOS-HIV scale is a 35-item measure of health related quality of life (QOL) questionnaire which assesses 10 dimensions of health (general health perceptions, pain, physical functioning, role functioning, social functioning, mental health, energy/fatifue, cognitive function, health distress and QOL), as well as a single item to assess health transition. In addition to these subscales, a Physical Health Summary score (PHS) and a Mental Health Summary score (MHS) is calculated using a method where the summary scores are transformed to a standardized scale with a norm of 50 and a standard deviation of 10 in the sample in which the summary scores were developed. The subscales of the MOS-HIV are scored as summed rating scales ranging from a minimum of 0, to a maximum of 100, where higher scores indicate better health.
Time Frame: Week 4 Follow-up
Population: Analyses were not performed due to too few participants.
Arm/Group | Raltegravir + 2 NRTIs | NNRTI + 2 NRTIs | PI + 2 NRTIs
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Depression, Anxiety, and Stress Scale (DASS-21)
Description: DASS-21 is comprised of questionnaires for three separate scales measuring Depression, Anxiety and Stress. The depression scale is scored by summing the responses of each question, multiplying by 2 and then scoring on a scale ranging from a minimum of 0 to a maximum of 28+, with higher scores indicating greater severity. The anxiety scale is scored by summing the responses of each question, multiplying by 2 and then scoring on a scale ranging from a minimum of 0 to a maximum of 20+, with higher scores indicating greater severity. The stress scale is scored by summing the responses of each question, multiplying by 2 and then scoring on a scale ranging from a minimum of 0 to a maximum of 37+, with higher scores indicating greater severity.
Time Frame: Baseline and Week 4 Follow-up
Population: Analyses were not performed due to too few participants.
Arm/Group | Raltegravir + 2 NRTIs | NNRTI + 2 NRTIs | PI + 2 NRTIs
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in HIV Symptom Index (HIV-SI)
Description: HIV-SI measures the frequency and level of bothersome HIV and HIV treatment-related symptoms, including nervous symptoms (dizziness, somnolence, trouble remembering), gastrointestinal symptoms (nausea, gas/bloating, diarrhea) and pain (hand/foot, muscle/joint). The 20-item questionnaire asks whether respondents experienced any one of these symptoms within the past 4 weeks, and if they did, what the relative level of bother for each symptom was, based on a 5-point Likert scale. The maximum sum of scores is 80; the minimum is 0; with a higher score indicating greater symptom distress.
Time Frame: Baseline and Week 4 Follow-up
Population: Analyses were not performed due to too few participants.
Arm/Group | Raltegravir + 2 NRTIs | NNRTI + 2 NRTIs | PI + 2 NRTIs
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: DLQI is a 10-question dermatology-specific QOL questionnaire, which is calculated by summing the score of each question, resulting in a maximum of 30, and a minimum of 0. Higher scores mean the QOL is more impaired.
Time Frame: Baseline and Week 4 Follow-up
Population: Analyses were not performed due to too few participants.
Arm/Group | Raltegravir + 2 NRTIs | NNRTI + 2 NRTIs | PI + 2 NRTIs
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days following end of the study's observation period
Arm/Group | Raltegravir + 2 NRTIs | NNRTI + 2 NRTIs | PI + 2 NRTIs
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/21 | 0/6
Other Adverse Events (participants affected / at risk) | 0/36 | 0/21 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes